CLINICAL TRIAL: NCT06529939
Title: The Effects of Psilocybin on Shared Experience in Film Processing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Adrian Owen, Professor of Cognitive Neuroscience and Imaging, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OWENLAB01
Record Dates: First submitted 2024-07-18; First posted 2024-07-31 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-07

CONDITIONS: Disorders of Consciousness; Psychedelic Experiences
Keywords: Psilocybin; Functional Magnetic Resonance Imaging (fMRI); Cognition; Disorders of Consciousness; Film Processing; Healthy Volunteers
MeSH Terms: conditions — Consciousness Disorders | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psilocybin First (Experimental): Individuals in this arm will be given psilocybin for their first scanning session. For their second scanning session (at least two weeks later), they will receive the placebo.
  Interventions: Drug: Psilocybin; Other: Placebo
- Placebo First (Experimental): Individuals in this arm will be given the placebo for their first scanning session. For their second scanning session (at least two weeks later), they will receive psilocybin.
  Interventions: Drug: Psilocybin; Other: Placebo

INTERVENTIONS:
Drug: Psilocybin — Individuals will be given 15 milligrams (mg) of psilocybin orally, and will be asked to lay flat in a functional magnetic resonance imaging (fMRI) brain scanner. The following scans will be collected: anatomical and resting state; while they watch a scrambled film clip; while they watch an intact film clip; while they perform a mental imagery task; while they listen to two pieces of music.
  Participants will then be given two questionnaires: one assessing their overall plot comprehension, and the other asking about their experience in the scanner. They will then be asked to perform a series of visual illusions tasks, and following, play a variety of web-based games assessing their cognitive function. After this, they will be interviewed by one of the study researchers about their overall experience before/during/after the scan.
Other: Placebo — Individuals will be given a placebo orally, and will be asked to lay flat in a functional magnetic resonance imaging (fMRI) scanner. The following scans will be collected: anatomical and resting state; while they watch a scrambled film clip; while they watch an intact film clip; while they perform a mental imagery task; while they listen to two pieces of music.
  Participants will then be given two questionnaires: one assessing their overall plot comprehension, and the other asking about their experience in the scanner. They will then be asked to perform a series of visual illusions tasks, and following, play a variety of web-based games assessing their cognitive function. After this, they will be interviewed by one of the study researchers about their overall experience before/during/after the scan.

SUMMARY:
The goal of this clinical trial is to learn whether certain methods of detecting awareness in vegetative or minimally conscious patients (using neuroimaging) are sensitive to the effects of psilocybin (a psychedelic drug). One of these methods includes scanning peoples' brains while they watch a film. When different individuals watch a film, their brains become synchronized with each other as they watch the plot unfold. Most importantly, if a seemingly unconscious patient also shows the same brain-synchronization, it means they might actually be conscious and aware.

To approach this goal, the investigators will be carrying out this trial in healthy volunteers. This will help better understand whether psilocybin may be a potential treatment for restoring awareness in these patients. The main questions it aims to answer are:

* Does psilocybin enhance or diminish brain synchrony during a film?
* Do changes in brain synchrony reflect differences in each individual's conscious experience?

Participants will be asked to:

* Attend two brain scanning sessions and watch a series of film clips, perform a brief mental imagery task, and listen to music - once under a placebo, and once under psilocybin.
* Play a series of games that assess their cognition (memory, reasoning, planning, etc.).
* Perform a series of visual illusions tasks.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* Have access to an internet connection
* Be in good general health
* Be 19 years of age, or older
* Be willing to follow the study protocol

Exclusion Criteria:

The following people will be excluded from the study. Those who:

* Are unable to read English
* Have high blood pressure
* Are pregnant (determined by a urine pregnancy test at in-person screening)
* Are not using effective methods of contraception with their partner(s) (e.g. oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine coil, intrauterine device, tubal ligation, or barrier method)
* Are taking chronic administration of tricyclic antidepressants and/or lithium
* Are taking acute administration of serotonin reuptake inhibitors
* Are currently using the antipsychotic medication haloperidol
* Are currently using monoamine oxidase inhibitors
* Have any current or past history of meeting the Diagnostic and Statistical Manual of Mental Illnesses (DSM-V) criteria for schizophrenia, bipolar I, bipolar II, or psychotic symptoms
* Have any first or second-degree relatives with history of above disorders/symptoms
* Have any other diagnosed and/or extreme psychiatric disorders, such as anxiety, depression, post-traumatic stress disorder (PTSD), addiction, obsessive-compulsive disorder (OCD), etc.
* Have any history of suicidal behaviour or current/recent suicidal ideation (determined by the Columbia-Suicide Severity Rating Scale [C-SSRS] at in-person screening)

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Intersubject Correlation (ISC) | Through study completion, an average of 2 weeks. ISC for each drug/task condition is computed and analyzed following second scan (from neuroimaging data).
  The degree to which different participants' brain activity is correlated with one another (or synchronized) across the time-course of an in-scanner task (e.g. during a resting state, while watching film clips, while listening to music, etc.). Higher ISC scores indicate greater brain synchronization between individuals (minimum value=0, indicating no ISC/synchronization).
Interpretive Phenomenological Analysis | Through study completion, an average of 2 weeks. Analyzed following second scan (from interview data).
  An analysis of the different themes that emerge (e.g. "feeling joy") when interviewing participants about their experience under the placebo or psilocybin. These themes will be correlated against ISC scores for each drug condition. Not scored on any scale; each theme's prevalence will be reported as a ratio and/or percentage.

SECONDARY OUTCOMES:
Short-Term Memory | Through study completion, an average of 2 weeks. Analyzed following second scan (from Creyos cognitive scores).
  An assessment of the short-term memory abilities of each participant. These scores are computed by the Creyos online cognitive testing platform, from each participants' performance on the suite of web-based games (which assess memory, spatial/verbal reasoning, planning, and concentration). Data will likely be reported as a normalized score with no min/max value (higher scores will indicate a better outcome).
Verbal Reasoning | Through study completion, an average of 2 weeks. Analyzed following second scan (from Creyos cognitive scores).
  An assessment of the verbal reasoning abilities of each participant. These scores are computed by the Creyos online cognitive testing platform, from each participants' performance on the suite of web-based games (which assess memory, spatial/verbal reasoning, planning, and concentration). Data will likely be reported as a normalized score with no min/max value (higher scores will indicate a better outcome).
Reasoning Skills | Through study completion, an average of 2 weeks. Analyzed following second scan (from Creyos cognitive scores).
  An assessment of the logical reasoning skills of each participant. These scores are computed by the Creyos online cognitive testing platform, from each participants' performance on the suite of web-based games (which assess memory, spatial/verbal reasoning, planning, and concentration). Data will likely be reported as a normalized score with no min/max value (higher scores will indicate a better outcome).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott G, Carhart-Harris RL. Psychedelics as a treatment for disorders of consciousness. Neurosci Conscious. 2019 Apr 21;2019(1):niz003. doi: 10.1093/nc/niz003. eCollection 2019. PMID 31024740
- [Background] Schartner MM, Carhart-Harris RL, Barrett AB, Seth AK, Muthukumaraswamy SD. Increased spontaneous MEG signal diversity for psychoactive doses of ketamine, LSD and psilocybin. Sci Rep. 2017 Apr 19;7:46421. doi: 10.1038/srep46421. PMID 28422113
- [Background] Hasson U, Landesman O, Knappmeyer B, Vallines I, Rubin N, Heeger DJ. Neurocinematics: The neuroscience of film. Projections. 2008;2(1):1-26.
- [Background] Naci L, Cusack R, Anello M, Owen AM. A common neural code for similar conscious experiences in different individuals. Proc Natl Acad Sci U S A. 2014 Sep 30;111(39):14277-82. doi: 10.1073/pnas.1407007111. Epub 2014 Sep 15. PMID 25225384
- [Background] Naci L, Sinai L, Owen AM. Detecting and interpreting conscious experiences in behaviorally non-responsive patients. Neuroimage. 2017 Jan 15;145(Pt B):304-313. doi: 10.1016/j.neuroimage.2015.11.059. Epub 2015 Dec 8. PMID 26679327